CLINICAL TRIAL: NCT04258319
Title: Sub-Hertz Analysis of Viscoelasticity of Limbs in Patients With Lymphedema
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Antonio J. Forte, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-005276
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: The unaffected arm will be used to serve as control for the affected extremity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Affected (Lymphedema) (Experimental): Subjects affected lymphedema extremity will have elastic and viscoelastic parameters collected by ultrasound procedure
  Interventions: Diagnostic Test: Ultrasound Procedure
- Unaffected (Control) (Active Comparator): Subjects unaffected extremity will have elastic and viscoelastic parameters collected by ultrasound procedure
  Interventions: Diagnostic Test: Ultrasound Procedure

INTERVENTIONS:
Diagnostic Test: Ultrasound Procedure — Ultrasound technique that uses a compression device integrated with ultrasound imaging to perform in vivo ramp-and-hold uniaxial creep-like test on upper extremity lymphedema (UEL) in vivo.

SUMMARY:
Researchers are trying to validate the use of ultrasound sub-hertz analysis of viscoelastisty (SAVE) method to monitor tissue-fluid dynamics and stage disease severity in patients diagnosed with lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Ability to provide written consent
* Has been diagnosed with Lymphedema

Exclusion Criteria:

* Under the age of 18 years old
* Inability to provide written consent
* Previous lymphovenous bypass or lymph node transfer surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Viscoelasticity parameters with lymphedema as obtained using the SAVE method | Baseline
  Defined as the difference in viscoelastic parameters between the arm affected with lymphedema and the unaffected extremity (affected minus unaffected) using the sub-hertz analysis of viscoelasticity method

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Forte, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No